CLINICAL TRIAL: NCT00820547
Title: Phase II Study Evaluating the Efficacy and Tolerance of Bevacizumab (Avastin) in HER2- Inflammatory Breast Cancer
Brief Title: Efficacy and Tolerance Study of Bevacizumab in Her2- Inflammatory Breast Cancer Patients
Acronym: Beverly1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACS09 UC-0140/0802; UNICANCER-PACS-09-0802 (Other: Internal Id Number); 2008-001807-53 (EudraCT Number)
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Breast Neoplasms, Male | interventions — Bevacizumab; Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (FEC / Docetaxel) + Bevacizumab (Experimental): Neoadjuvant treatment: 4 cycles FEC + Bevacizumab followed by 4 cycles Docetaxel + Bevacizumab Adjuvant: Bevacizumab for 1 year
  Interventions: Biological: bevacizumab; Drug: cyclophosphamide; Drug: docetaxel; Drug: epirubicin hydrochloride; Drug: fluorouracil

INTERVENTIONS:
Biological: bevacizumab — During neoadjuvant phase: 15 mg/kg, d1 q3w, 8 cycles During adjuvant phase:15 mg/kg, d1 q3w, 10 cycles
Drug: cyclophosphamide — Neoadjuvant: 500 mg/m2 d1 q3w, 4 cycles
Drug: docetaxel — Neoadjuvant: 100 mg/m2 q3w, 4 cycles
Drug: epirubicin hydrochloride — Neoadjuvant: 100 mg/m2, d1 q3w, 4 cycles
Drug: fluorouracil — Neoadjuvant: 500 mg/m2, d1 q3w, 4 cycles

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab and combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving bevacizumab and radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying giving bevacizumab together with chemotherapy before surgery and bevacizumab and radiation therapy after surgery to see how well it works in treating patients with inflammatory breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the complete histological response rate in patients with inflammatory HER2-negative breast cancer treated with bevacizumab and concurrent chemotherapy followed by bevacizumab and concurrent hormonal therapy after surgery and radiotherapy.

Secondary

* Evaluate the progression-fee and overall survival of these patients at 3 and 5 years.
* Evaluate the tolerance of bevacizumab in these patients.
* Assess circulating metastatic disease before, during, and after treatment.
* Assess circulating endothelial cells before, during, and after treatment.
* Assess predictive factors of response by genomic and proteomic studies on frozen tumor samples and fluid samples (i.e., serum and plasma).

OUTLINE: This is a multicenter study.

* Neoadjuvant induction therapy:

  * Courses 1-4: Patients receive bevacizumab IV over 30-90 minutes, fluorouracil IV, epirubicin hydrochloride IV over 10 minutes, and cyclophosphamide IV over 5 minutes on day 1.
  * Courses 5-8: Patients receive bevacizumab IV over 30-90 minutes and docetaxel IV over 1 hour on day 1.

Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

* Surgery: Patients undergo surgery 4-6 weeks after completion of bevacizumab.
* Adjuvant therapy: Beginning 2-4 weeks after surgery, patients undergo radiotherapy for 6 weeks. Patients also receive bevacizumab IV over 30-90 minutes beginning 2-4 weeks after surgery, during the radiotherapy period. Treatment with bevacizumab repeats every 3 weeks for 30 weeks in the absence of disease progression or unacceptable toxicity. Patients who are estrogen receptor- or progesterone receptor-positive (≥ 10% by IHC) receive the following concurrent hormonal therapy beginning in week 7:

  * Premenopausal patients: Patients receive tamoxifen citrate for 5 years.
  * Postmenopausal patients: Patients receive aromatase-inhibitor therapy (or tamoxifen citrate if unable to tolerate anti-aromatase therapy) for 5 years.
  * Perimenopausal patients: Patients receive tamoxifen citrate for 2-3 years and aromatase-inhibitor therapy for 2-3 years OR tamoxifen citrate for 5 years followed by aromatase-inhibitor therapy for 2-3 years (if follicle-stimulating hormone > 30 IU/L and/or estradiol < 30 ng/L).

After completion of study treatment, patients are followed for at least 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed inflammatory breast cancer, meeting 1 of the following staging criteria:

  * T4d, any N (AJCC stage IIIB or IIIC)
  * Gustave-Roussy Institute (IGR) classification Poussee evolutirie (PEV; measures tumor growth over time) 2

    * PEV 2: tumor with underlying breast tissue, especially skin, that is affected by subacute inflammation and edema involving < ½ of breast surface
  * IGR classification PEV 3

    * PEV 3: acute or subacute inflammation and edema involving > ½ of breast surface
  * Biopsy-confirmed presence of tumor embolism in surface lymph nodes
* HER2-negative (HER2 0 or 1+, or HER2 2+ by IHC if FISH-negative allowed)
* No metastatic disease
* No non-inflammatory breast cancer with edema, ulceration, or satellite skin nodules
* No bilateral breast cancer
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Any menopausal status allowed
* WHO performance status 0-2
* Life expectancy ≥3 months
* LVEF normal by ECHO
* ANC >1.5 x 10^9/L
* Platelet count >100 x 10^9/L
* INR ≤1.5 (except for patients on prophylactic anticoagulants)
* aPTT ≤1.5 times upper limit of normal (ULN)
* Total bilirubin normal
* SGOT and SGPT ≤1.25 times ULN
* Alkaline phosphatase ≤2.5 times ULN
* Creatinine clearance ≥60 mL/min
* Proteinuria <2+ or 24-hour urine protein ≤1 g
* No unhealed wound, stomach ulcer, or bone fracture
* No history of thrombotic or hemorrhagic disorders
* No significant cardiovascular disease including the following:

  * Cerebrovascular accident within the past 6 months
  * Unstable angina
  * Cardiac failure
  * Myocardial infarction
  * Arrhythmia requiring treatment
* No uncontrolled hypertension (i.e., systolic BP >150 mm Hg and/or diastolic BP >100 mm Hg)
* No other active infection or serious illness that would preclude patient from receiving study treatment
* No hypersensitivity to any active products or excipients of study drugs
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No social or psychologic reasons that would prevent study compliance or follow-up
* No patients who are incarcerated or on probation

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or hormonal therapy for this disease
* More than 4 weeks since prior surgery (diagnostic biopsy or installation of implant allowed)
* More than 10 days since prior chronic non-inflammatory steroids (e.g., acetylsalicylic acid >325 mg/day) or platelet anticoagulation treatment (e.g., dipyridamole, ticlopidine, clodiprogel, cilostazol)
* More than 10 days since prior oral or parenteral anticoagulant or thrombolytic drugs (preventative thrombolytic drugs allowed)
* No concurrent participation in another experimental clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Complete histologic response rate | Post surgery

SECONDARY OUTCOMES:
Progression-free survival | 3 and 5 years
Overall survival | 3 and 5 years
Toxicity as assessed by CTCAE v3.0 | 3 and 5 years
Predictive factors of response to bevacizumab | 3 and 5 years
Circulating peripheral cells (circulating endothelial and tumor cells): correlation of initial rate and association with histological response after surgery | Post-surgery
Genomic and proteomic analyses and correlation with histologic response | Post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Viens, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (28):
- France (28):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - CMC Les Ormeaux, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Hospitalier General Andre Boulloche, Montbéliard
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Hopital, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - CRLCC Nantes - Atlantique, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported under the following conditions: the data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Bertucci F, Fekih M, Autret A, Petit T, Dalenc F, Levy C, Romieu G, Bonneterre J, Ferrero JM, Kerbrat P, Soulie P, Mouret-Reynier MA, Bachelot T, Lerebours F, Eymard JC, Deblock M, Lortholary A, Hardy-Bessard AC, Barthelemy P, Bonnefoi H, Charafe-Jauffret E, Bidard FC, Viens P, Lemonnier J, Pierga JY. Bevacizumab plus neoadjuvant chemotherapy in patients with HER2-negative inflammatory breast cancer (BEVERLY-1): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2016 May;17(5):600-11. doi: 10.1016/S1470-2045(16)00011-5. Epub 2016 Mar 28. PMID 27032301
- See also: Abstract results — https://www.ncbi.nlm.nih.gov/pubmed/27032301